CLINICAL TRIAL: NCT07005141
Title: iHub no Tratamento de Aneurismas ilíacos: Avaliação da Segurança, Desempenho e Eficácia.
Brief Title: iHub Stent-Graft for Iliac Artery Aneurysms: Safety, Performance, and Effectiveness Study
Acronym: TriHub
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Archo Medical S.A (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.A.1-PRT-SRE-005.02
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Iliac Aneurysm; Aortic Aneurysm, Abdominal
Keywords: iliac aneurysm; iHub; stentgraft system; endovascular treatment; abdominal aortic aneurysm; EVAR
MeSH Terms: conditions — Iliac Aneurysm; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovascular Implant of iHub Iliac Stent-Graft for Treatment of Iliac Artery Aneurysms (Experimental): Eligible participants with an iliac artery aneurysm, or aneurysms of the iliac arteries, who have iliac/femoral access compatible with the delivery systems, and a previously implanted or concurrently implanted bifurcated aortic stent-graft with branch diameters between 14 and 16 mm, will undergo endovascular surgery for aneurysm treatment using the iHub device
  Interventions: Device: Endovascular Iliac Branch Stent-Graft Implantation

INTERVENTIONS:
Device: Endovascular Iliac Branch Stent-Graft Implantation — Implantation of a self-expanding dual-lumen iliac branch stent-graft designed to treat iliac artery aneurysms while preserving perfusion to the internal iliac artery. The device enables connection to bridging stent-grafts directed to both the internal and external iliac arteries. It is compatible with previously implanted or concurrently implanted bifurcated aortic stent-grafts with branch diameters between 14 and 16 mm. The stent-graft is delivered endovascularly using a low-profile catheter-based system under fluoroscopic guidance. Once in position, the device is deployed via a controlled pull-back release mechanism. Radiopaque markers assist in precise alignment and facilitate the placement of bridging components.
  Other Names: Implantation of an Endovascular Iliac Branch Stent-Graft for Iliac Aneurysm Repair

SUMMARY:
The goal of this clinical trial is to evaluate the safety, performance, and Preliminary effectiveness of the iHub endoprosthesis system in treating iliac artery aneurysms in adult patients requiring endovascular repair. The study population includes both male and female adults over 18 years of age who meet the inclusion criteria for endovascular treatment of iliac artery aneurysms.

The main questions it aims to answer are:

Is the iHub stent-graft system safe for use in patients with iliac artery aneurysms? Does the iHub system demonstrate adequate technical performance and sustained patency over a 12-month follow-up period? Participants will undergo a minimally invasive endovascular procedure to implant the iHub endoprosthesis system. The device is designed to preserve internal iliac artery flow while excluding the aneurysmal segment.

Participants will:

Undergo pre-screening evaluations including clinical examination, laboratory tests, and imaging (CT angiography and ultrasound).

Undergo endovascular implantation of the iHub device. Attend follow-up visits at 30, 90, 180, and 360 days post-implant to assess clinical outcomes and device performance.

DETAILED DESCRIPTION:
This study investigates the first-in-human use of the iHub Stent-Graft System, a vascular endoprosthesis developed to treat aneurysms in the iliac arteries with an emphasis on preserving internal iliac artery (IIA) perfusion and minimizing complications associated with pelvic ischemia. The iHub device represents an innovation in the treatment of complex aortoiliac aneurysms by offering a novel anatomical configuration and deployment strategy.

Scientific Background and Rationale

Iliac artery aneurysms (IAA), particularly those involving the common iliac artery (CIA) and extending to the internal iliac artery, pose a treatment challenge due to the anatomical and hemodynamic complexity of the pelvic vasculature. The interruption of flow to the IIA has been associated with postoperative complications such as buttock claudication, sexual dysfunction, and colonic ischemia. Therefore, preserving the IIA during endovascular aneurysm repair (EVAR) is a priority in complex iliac anatomy.

The iHub device is designed to offer a modular and flexible approach to treating iliac aneurysms, incorporating branch preservation without requiring total exclusion of the internal iliac circulation. The study addresses a significant unmet clinical need, especially in patients who are not good candidates for conventional bifurcated aortic endografts or hybrid procedures.

Device Description

The iHub stent-graft is a low-profile device delivered via catheter for the treatment of Iliac Artery Aneurysm (IAA). The device is designed to exclude common iliac artery aneurysms while simultaneously preserving internal iliac artery perfusion.

The stent-graft consists of a single tubular component made of a self-expanding nitinol stent covered with an ePTFE film. Internally, this polymeric tube divides into two smaller tubes, measuring 9 ± 1 mm and 7 ± 1 mm in diameter, each 20 mm in length. This configuration allows the stent-graft to connect, via bridging stent-grafts, to both the internal and external iliac arteries.

For implantation, the stent-graft is compressed within a delivery system (introducer catheter), which transports the device to the target site. Once released, the stent-graft expands to its nominal diameter. The stent-grafts are manufactured in a size suitable for implantation into a main endograft branch with diameters ranging from 14 mm to 16 mm.

The stent-graft is preloaded into an introducer system, and once it reaches the intended implantation site, the device is released. During positioning, a pull-back maneuver is used to deploy the stent-graft under fluoroscopic guidance. Immediately afterward, the system's inner mandrel is removed, and the catheter then functions as an introducer sheath through which the external iliac bridging stent-graft is delivered.

The delivery system is preassembled and single-use, sterilized via ethylene oxide (EO) and validated according to ISO 11135, with sterile barrier packaging conforming to ISO 11607-1 and 11607-2.

Objectives and Expected Outcomes

To evaluate the performance of the iHub stent-graft in patients with iliac artery aneurysms. The specific objectives are:

I. To assess the safety of the iHub iliac stent-graft at 30, 90, 180, and 360 days post-implantation.

II. To evaluate the accuracy of the iHub stent-graft deployment at the intended anatomical location.

III. To assess the effectiveness of the iHub stent-graft in excluding the iliac artery aneurysm.

Primary objective is the absence of serious adverse events related to the device within 30 days following the endovascular procedure.

The secundary objective is to evaluate the performance of the iHub Stent-Graft in patients with Iliac Artery Aneurysms. Performance is defined as:

1. Successful implantation of the stent-graft device in one or both iliac branches and exclusion of the common iliac artery aneurysm.
2. Absence of Type I, III, and IV endoleaks during the 30-day follow-up period.
3. Incidence of serious adverse events at 90, 180, and 360 days post-implantation.

Study Design and Monitoring

This is a prospective, multicenter, first-in-human, interventional clinical investigation. Patients will undergo treatment at a qualified vascular surgery center under the oversight of a designated principal investigator (PI). The surgical team will follow a defined implant protocol, including preoperative imaging, device sizing, and procedural technique as outlined in the investigator brochure.

Monitoring of safety parameters will occur at regular intervals post-implantation through structured follow-up visits. Each follow-up includes standardized physical exams, imaging studies (ultrasound, RX and CT angiography), and laboratory testing to assess renal function.

All clinical events, including adverse events and serious adverse events (SAEs), will be tracked and categorized using standard definitions provided by ISO 14155 and Good Clinical Practice (GCP) guidelines. Data management, event adjudication, and protocol compliance monitoring will be performed by the sponsor and independent clinical monitors.

Risk Assessment and Patient Safety

The potential risks of this study include access failures, device migration, endoleaks, device fracture or infection, and cardiac, pulmonary, renal, neurological, genitourinary, sexual, thrombotic, inflammatory, anesthetic-related complications, and death. To mitigate these risks, robust qualification tests were performed on the device, quality control measures were applied during manufacturing, and experienced investigators in endovascular procedures were selected. All study personnel will receive detailed training on the protocol, device usage, and participant follow-up. A follow-up schedule, well-defined inclusion/exclusion criteria, and continuous monitoring of data and adverse events will be implemented. Safety and performance outcomes will be shared with the investigative centers throughout the study.

Ethical Considerations

The protocol was developed in compliance with ISO 14155:2020 for clinical investigation of medical devices for human subjects and follows Brazilian regulations including RDC 751/2022 , CNS 466/12 and RDC 837/2023. Ethical approval will be obtained from a local Research Ethics Committee (Comitê de Ética em Pesquisa - CEP), and all patients will sign informed consent prior to enrollment.

The consent process emphasizes voluntariness, right to withdraw at any time, and clarification of potential risks, benefits, and alternative treatments. The study complies with the ethical principles outlined in the Declaration of Helsinki.

Data Analysis and Reporting

Quantitative analysis will be performed on both safety and performance endpoints. Descriptive statistics will be used to summarize patient demographics, procedural metrics, and adverse event frequencies. Device performance will be assessed through imaging-based outcomes, including patency of the branch, endoleak classification, and aneurysm exclusion.

Any need for secondary intervention, as well as clinical symptoms such as claudication or pelvic ischemia, will be recorded. Data will be analyzed at key time points: baseline, hospital discharge, and at 90, 180, and 360 days post-procedure.

Significance and Future Directions

This study is intended to provide foundational data for future regulatory submissions. It will help determine the real-world utility and safety profile of the iHub system in the treatment of iliac aneurysms requiring internal iliac artery preservation.

If successful, the iHub may represent a valuable tool in the endovascular armamentarium, providing a lower-profile, flexible option for patients with complex iliac anatomy.

ELIGIBILITY:
Inclusion Criteria: Sign the Informed Consent Form (ICF); Are ≥ 18 years of age;

Meet at least one of the following criteria for iliac artery aneurysm:

1. Common iliac artery aneurysm ≥ 25 mm in diameter;
2. Aneurysm growth of 5 mm or more within the last six months;
3. Maximum aneurysm diameter exceeds 1 to 1.5 times the normal arterial segment diameter, that is ≥ 25 mm maximum diameter;
4. Saccular aneurysm greater than 20 mm;
5. Abdominal aortic aneurysm with extension into the common iliac arteries of less than 20 mm;

Have a previously implanted aorto-bi-iliac stent-graft with branch diameter between 14 and 16 mm;

Have iliac/femoral access vessel morphology compatible with vascular access techniques, placement systems, devices, and/or accessories;

Are classified as ASA physical status I to III. ASA IV patients may be included if their life expectancy is greater than one year;

Are able and willing to comply with follow-up requirements during the 360-day post-implant period.

-

Exclusion Criteria: Pregnant women, women of childbearing potential, or breastfeeding women;

A dissection, rupture, or complex vascular lesion due to trauma;

Need for emergency surgery;

Contraindication to angiography;

Diffuse atherosclerotic disease in any common iliac artery reducing its diameter to < 4 mm;

Congenital abnormalities where stent placement would obstruct a major artery. Such abnormalities must be assessed prior to treatment;

Unstable angina;

Class III obesity (BMI ≥ 40 kg/m²) or other clinical conditions that severely limit radiographic visualization of the aorta;

Connective tissue disease (e.g., Marfan or Ehlers-Danlos syndrome);

Hypercoagulable state;

Contraindication to anticoagulation therapy;

Acute or chronic renal insufficiency (serum creatinine > 2.0 mg/dL);

Life expectancy of less than one year;

Presence of a systemic infection that could increase the risk of endovascular device infection;

Known sensitivity or allergy to device materials: expanded polytetrafluoroethylene (ePTFE), fluorinated ethylene propylene (FEP), or nickel-titanium (Nitinol).

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Absence of serious adverse events related to the device in the first month after the procedure | Within 30 days after implantation
  Absence of serious adverse events related to the investigational device within 30 days after implantation. These events include, but are not limited to, stent-graft migration, vessel dissection, stent-graft obstruction, occlusion of collateral vessels, type I, III, and IV endoleaks, aneurysm rupture, and intraoperative mortality.

SECONDARY OUTCOMES:
Absence of surgical conversion during the follow-up period from 3 to 12 months and device performance | Follow-up period from 3 to 12 months
  Absence of surgical conversion should occur during the follow-up period from 3 to 12 months and absence of leaks (endoleaks).Besides absence os incidence of serious adverse events. The study also aims to demonstrate successful delivery system positioning and accurate deployment of the stent-graft at the intended anatomical site.

CONTACTS AND LOCATIONS:
Overall Officials: Grace C Mulatti, PI, Principal Investigator — Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo- FMUSP
Locations (2):
- Brazil (2):
  - Hospital Baía Sul S/A, Florianópolis, Santa Catarina
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo - HCFMUSP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) that underlie the results reported in this study will be shared, including:
  Demographic data (e.g., age, sex, baseline comorbidities)
  Epidemiological data relevant to the target population affected by aortoiliac aneurysms
  Procedural data related to technical success, including device deployment, patency, and procedural complications
  Clinical outcomes used to define primary and secondary success, including imaging follow-up and adverse events
  All collected IPD that support the assessment of primary and secondary endpoints, including freedom from endoleaks, graft patency, reintervention rates, and overall survival
  Technical success data, including successful access, delivery, deployment, and placement of the iHub device as per protocol
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available beginning 12 months after the final publication of the primary results and will remain accessible for at least 5 years.
Access Criteria: Data will be available to qualified researchers upon reasonable request, subject to approval by the sponsor and compliance with data privacy regulations and applicable ethical standards.
URL: https://archomedical.com